CLINICAL TRIAL: NCT05526313
Title: Single-center, Dose-escalation Phase I Tolerability, Safety, Pharmacokinetics and Efficacy of Purinostat Mesylate (PM) for Injection in the Treatment of Relapsed or Refractory B Cell-related Tumor-predominant Hematologic Tumors Clinical Trials for Pharmacodynamic Evaluation
Brief Title: Study of Purinostat Mesylate for Injection in the Treatment of Relapsed or Refractory B Cell-related Tumor-predominant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GZ2018-001-1.0
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Large B Cell Lymphoma，DLBCL
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 1.2mg/m^2 (Experimental)
  Interventions: Drug: Purinostat Mesylate 1.2mg/m^2
- 2.4mg/m^2 (Experimental)
  Interventions: Drug: Purinostat Mesylate 2.4mg/m^2
- 4.0mg/m^2 (Experimental)
  Interventions: Drug: Purinostat Mesylate 4.0mg/m^2
- 6.0mg/m^2 (Experimental)
  Interventions: Drug: Purinostat Mesylate 6.0mg/m^2
- 8.4mg/m^2 (Experimental)
  Interventions: Drug: Purinostat Mesylate 8.4mg/m^2
- 11.2mg/m^2 (Experimental)
  Interventions: Drug: Purinostat Mesylate 11.2mg/m^2
- 15mg/m^2 (Experimental)
  Interventions: Drug: Purinostat Mesylate 15mg/m^2

INTERVENTIONS:
Drug: Purinostat Mesylate 1.2mg/m^2 — 1 case,The starting dose,Take the medicine once on D1, D8, D11, D15.
  Arms: 1.2mg/m^2
Drug: Purinostat Mesylate 2.4mg/m^2 — Take the medicine once on D1, D8, D11, D15.
  Arms: 2.4mg/m^2
Drug: Purinostat Mesylate 4.0mg/m^2 — Take the medicine once on D1, D8, D11, D15.
  Arms: 4.0mg/m^2
Drug: Purinostat Mesylate 6.0mg/m^2 — Take the medicine once on D1, D8, D11, D15.
  Arms: 6.0mg/m^2
Drug: Purinostat Mesylate 8.4mg/m^2 — Take the medicine once on D1, D8, D11, D15.
  Arms: 8.4mg/m^2
Drug: Purinostat Mesylate 11.2mg/m^2 — Take the medicine once on D1, D8, D11, D15.
  Arms: 11.2mg/m^2
Drug: Purinostat Mesylate 15mg/m^2 — Take the medicine once on D1, D8, D11, D15.
  Arms: 15mg/m^2

SUMMARY:
Purinostat mesylate for injection (PM) was the novel and highly potent Class I a and IIb HDAC-selective inhibitors. The results of regular blood sampling analysis of the mouse B-cell lymphoma model induced by ighmyc transgenic mice showed that the treatment of PM in each group reduced the proportion of peripheral blood tumor cells in mice. Therefore, PM has the potential to treat diffuse large B cell lymphoma.

The results of in vitro enzymatic activity screening showed that PM has high inhibitory activity on HDAC tumors (including HDAC1, 2, 3, 8 subtypes) and type II HDACs (including HDAC6, 10 isoforms), which are closely related to tumors in the HDAC family. Therefore, the results of in vitro enzyme activity screening showed that the IC50 values of PM for inhibiting HDAC1, HDAC2, HDAC3, HDAC8, HDAC6, and HDAC10 subtypes of HDAC class I and HDAC class IIb were 0.81, 1.4, 1.7, 3.8, 11.5, and 11 nM, respectively. However, the inhibitory activity of HDAC IIa and HDAC IV enzymes was low, and its IC50 values for HDAC4, HDAC5, HDAC7, HDAC9, and HDAC11 subtypes of HDAC IIa and HDAC IV were 1072, 426, 590, 622, and 3349 nM, respectively. These data means PM exist high selectivity for tumor-associated HDAC class I and HDAC IIb.

Compared with the blank control group, the body weight of the tumor-bearing animals in each dose of PM group did not decrease seriously during the treatment process, and the animals were in good condition during the whole experiment, indicating that the PM is efficacy and safe.

During the course of the experiment, the tumor cell population (GFP+, B220+) in the blood of the animals basically regressed after treatment with Prilistat hydrochloride.

Research purposes:

Main purpose:

Observation of patients with relapsed or refractory hematological tumors (including but not limited to after standard therapy) mainly in patients with relapsed or refractory B cell-related tumors. Tolerability and safety of B-cell lymphoma, multiple myeloma, B-cell acute leukemia, T-cell lymphoma, T-cell acute leukemia) with disease progression or ineligible for standard therapy.

To observe the dose-limiting toxicity (DLT) in patients with relapsed or refractory B cell-related tumors and hematological tumors, and determine its maximum tolerated dose (MTD), which is the maximum tolerated dose (MTD). Phase II clinical dosing schedule provides the basis.

Secondary Purpose:

To evaluate the pharmacokinetic parameters of patients with relapsed or refractory B-cell-related tumors and hematological tumors after single and multiple intravenous infusions of priinostat mesylate for injection.

To evaluate the pharmacodynamics of patients with relapsed or refractory B cell-related tumors and hematological tumors after single and multiple intravenous infusions of priinostat mesylate for injection.

To preliminarily observe the efficacy of Priinostat mesylate for injection in the treatment of patients with relapsed or refractory hematological tumors, mainly patients with B cell-related tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 to 70 years old, gender is not limited;
* 2. Hematological tumors, including but not limited to B-cell lymphoma, multiple myeloma, B Cell acute leukemia, T-cell lymphoma, T-cell acute leukemia, and patients with disease progression, relapse, or ineligibility for standard regimen therapy after standard regimen therapy ;
* 3. Patients without serious organic lesions in the heart, lung, liver and kidney (LVEF (left ventricular ejection fraction >=50%; total bilirubin <=1.5×ULN; alanine aminotransferase (ALT) <=1.5×ULN; aspartate aminotransferase); (AST) <=1.5×ULN (; serum creatinine<=1.5×ULN or CCr>40mL/min);
* 4. Those without severe coagulation dysfunction (PT<=1.5×ULN, APTT<=1.5×ULN, TT<=1.5×ULN and FIB>=1.0 g/L);
* 5. Patients without severe hematopoietic dysfunction (absolute neutrophil value>=1.5×109/L, platelets >=75×109/L, hemoglobin>=80g/L), and no platelet, red blood cell, hemoglobin;
* 6. Patients received at least 4 weeks or more than 5 half-lives after the last antitumor treatment (chemotherapy, radiotherapy, biological therapy or immunotherapy) before enrollment;
* 7. Expected survival time>= 12 weeks;
* 8. ECOG score <=2 points;
* 9. Those who agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

* 1. The toxicity of previous anticancer therapy has not recovered to grade I or below, or has not fully recovered from previous surgery;
* 2. Those with severe heart, lung, liver, kidney, digestive system diseases and chronic diseases of vital organs
* 3. Pregnant or breastfeeding female patients, fertile female/male patients who refuse to use contraceptive measures during the trial;
* 4. A history of acute myocardial infarction, congestive heart failure, unstable angina pectoris, or stroke within 6 months before enrollment;
* 5. Patients with impaired cardiac function (ejection fraction <45% detected by echocardiography or complete left bundle branch block with ECG ST segment downshift >1 mm or T wave inversion in two or more channels; congenital ventricular or Atrial arrhythmia, clinically significant tachycardia (>100 beats/min), bradycardia (<50 beats/min), ECG QTc >450 ms (men), QTc >480 ms (women), or clinically significant cardiac Diseases (such as unstable angina, congestive heart failure, myocardial infarction within 6 months), etc.;
* 6. Those with central nervous system lymphoma/leukemia or mental disorders;
* 7. Have a history of organ transplantation;
* 8. Those with severe active infection;
* 9. Known severe hypersensitivity to the test drug and its excipients or HDAC inhibitors;
* 10. HCV antigen or antibody positive, HIV antigen or antibody positive, HBsAg positive, HBcAb positive and peripheral blood HBV DNA titer detection >=1×103 IU/mL;
* 11. Alcohol dependence or drug abusers;
* 12. Those who have participated in clinical trials of other drugs within the past 1 month;
* 13. The researchers conclud that there are other factors that are not suitable for participating in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Purinostat Mesylate Pharmacokinetics (PK)：Cmax | 72hours
  Estimation of maximum observed plasma concentration
Purinostat Mesylate Pharmacokinetics (PK)：Tmax | 72hours
  Estimation of time to reach Cmax
Purinostat Mesylate Pharmacokinetics (PK)：AUC0-72h | 72hours
  Estimation of AUC from time zero to the last measured time point
Purinostat Mesylate Pharmacokinetics (PK)：AUC0-∞ | 72hours
  Estimation of AUC from time zero extrapolated to infinity
Purinostat Mesylate Pharmacokinetics (PK)：MRT | 72hours
  Estimation of mean residence time
Purinostat Mesylate Pharmacokinetics (PK)：Vd | 72hours
  Estimation of apparent volume of distribution
Purinostat Mesylate Pharmacokinetics (PK)：t1/2 | 72hours
  Estimation of terminal elimination half-life
Purinostat Mesylate Pharmacokinetics (PK)：CLz/F | 72hours
  Estimation of clearance when dosed orally
Purinostat Mesylate Pharmacokinetics (PK)：Vz/F | 72hours
  Estimation of apparent volume of distribution when dosed orally
Purinostat Mesylate Pharmacokinetics (PK)：Ke | 72hours
  Estimation of the elimination rate constant of a drug in the body

CONTACTS AND LOCATIONS:
Overall Officials: Ting Niu, Doctor, Principal Investigator — West China Hospital; Yongsheng Wang, Doctor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No